CLINICAL TRIAL: NCT02650661
Title: A Randomized Controlled Trial of Smart Management Strategy for Health (SMASH) Program for Overcoming Cancer Crisis and Growing Positively in Cancer Survivors
Brief Title: Efficacy of a Smart Management Strategy for Health (SMASH) Program for Overcoming Cancer Crisis and Growing Positively
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Samsung Medical Center (Other); Asan Medical Center (Other); Ewha Womans University Mokdong Hospital (Other); National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Young Ho Yun, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: YHYun
Record Dates: First submitted 2015-10-01; First posted 2016-01-08 (Estimated); Last update posted 2018-10-19 (Actual); Status verified 2018-10

CONDITIONS: Breast Neoplasms; Lung Neoplasms; Colorectal Neoplasms; Stomach Neoplasms
Keywords: Cancer survivors
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Colorectal Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Online program & Health coaching (Experimental): This group is provided with "Online health management program", "Health coaching" and "Workshop".
  Interventions: Behavioral: Online health management program; Behavioral: Health coaching; Behavioral: Workshop
- Online program (Experimental): This group is provided with "Online health management program".
  Interventions: Behavioral: Online health management program
- Enhanced Usual Care (Active Comparator): This group is provided with "Standard health educational booklet".
  Interventions: Behavioral: Standard health educational booklet

INTERVENTIONS:
Behavioral: Online health management program — Web-based health management program designed according to SMASH strategy, which includes (i) Assessment, (ii) Acceptance, (iii) Preparation for change, (iv) Commitment, (v) Planning, (vi) Promoting environment, (vii) Execution, (viii) Feedback and Maintenance, and (ix) Core perspectives, for 6 months.
  The program consists of four areas: self-assessment, self-planning, self-learning, and self-monitoring. The learning session includes SMASH strategies and "10 Rules for Highly Effective Health Behavior".
  Other Names: "Healthing U"
  Arms: Online program; Online program & Health coaching
Behavioral: Health coaching — Personalized tele-coaching for 6 months by health coaches who were trained by the Smart Management and Coaching for Health (SMACH) program
  Arms: Online program & Health coaching
Behavioral: Workshop — Total three sessions are to be held at 3-, 5-, and 7-month after the initiation of the enrollment. Each session includes 30-minute health education, 1-hour health management strategy workshop, and 30-minute team coaching.
  Other Names: Group education
  Arms: Online program & Health coaching
Behavioral: Standard health educational booklet — Standard health educational booklets about "10 Rules for Highly Effective Health Behavior" that are organized according to the Trans-theoretical Model (TTM).
  Booklets are provided at 0-, 2-, and 4-month after the enrollment.
  Arms: Enhanced Usual Care

SUMMARY:
The purpose of this study is to evaluate the efficacy of the "Smart Management Strategy for Health (SMASH)" program, which is designed to help cancer patients overcome their cancer crisis proactively and grow positively.

DETAILED DESCRIPTION:
<Hypothesis> This study hypothesizes that the intervention being provided (SMASH program) will demonstrate improvements in cancer survivors' health management in the fields of (i) physical activity, body mass index, and positive growth, (ii) self-management strategies of health (SMASH Assessment Tool; SAT), (iii) overall physical, mental, social, spiritual health conditions and Quality of Life (QoL), and (iv) the execution and maintenance of health habits ("10 Rules for Highly Effective Health Behavior").

<Patient registry> Cancer survivors, who have just completed their cancer treatments (surgery, radiation, chemotherapy), will be recruited from five medical centers in Korea and randomly allocated to one of following three groups: 2 experiment groups and 1 attention control group. This recruitment process would start after the approval of protocol by the Institutional Review Board (IRB), and proceed through following steps: (i) the physician in charge confirms that the patient has finished his or her treatment and determines whether the patient is eligible to participate in the study by checking the recent (less than one year) results of the patient's basic medical exams (blood pressure, body temperature, heart rate, respiratory rate, weight, and height) and basic lab tests (blood chemistry, electrocardiogram, chest PA, complete blood count, liver function test, BUN/Cr), (ii) A nurse explains the purpose and method of the study to the patient, and asks to complete informed consent form, (iii) the patient who agrees for participation will complete a brief screening questionnaire (Godin's Leisure Time Exercise, weight/height, and PostTraumatic Growth Inventory(PTGI)), (iv) the patient meeting the criteria as determined by the screening questionnaire is asked to complete the baseline assessment questionnaire at home, (v) cases who finish the baseline assessment questionnaire and meet all criteria are considered study participants and are randomly assigned to one of the three study arms.

<Quality control (patient data)> This study assumes that patients who are directly referred to the study by collaborating physicians are valid cancer cases. Data collected from study participants on screening forms will be reviewed by researchers at the central institution for missing responses and inconsistencies.

<Sample size>

The sample size of 477 participants was based upon the following assumptions:

* a two-sided Type I error of 0.05
* drop-out rate of 10%
* an attainment of goal behavior of 5% in the active comparator arm and 20% in the experiment arm, and a power of 90% to detect a between-arm difference

<Statistical analysis plan > The primary endpoint was based on three-outcome composite achievement of PA, weight and PTGI score at 12 months. All analyses will be conducted on the basis of intention-to-treat. Arm differences at 3, 6, and 12 months in behavior change (physical activity, body mass index, posttraumatic growth) will be tested with logistic regression, controlling for the respective baseline values. Arm differences in levels of Mini Dietary Assessment Index (MDI), execution of health habits, SMASH Assessment Tool (SAT), Quality of Life (QoL), health condition, incurred medical expenses, incurred Complementary and Alternative Medicine (CAM) expenses will be explored using a mixed model that estimates the effect of SMASH program over time, which will correlate repeated observations on particular participants after adjustment for baseline scores.

ELIGIBILITY:
Inclusion Criteria:

* Aware of one's diagnosis of breast, lung, colorectal or gastric cancer
* less than 2 months has passed since one's completion of primary cancer treatment (including surgery, radiation, or chemotherapy)
* Performs poorly at baseline on at least one goal behavior, which includes the followings:

  (i) moderate exercise ≥150 min/week or strenuous exercise ≥75 min/week (*exception: ≥12.5 MET-hr/week for lung cancer patients) (ii) BMI within normal range (18.5-22.9) (*exception: ≥18.5 for lung cancer patients) (iii) Posttraumatic Growth Inventory (PTGI) score ≥72

Exclusion Criteria:

* Inability to speak or write Korean
* Medical conditions that would limit adherence to an unsupervised health management program (as confirmed by their referring physician; e.g. major depression, dyspnea)
* Currently pregnant or planning to be within the next year

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 394 (Actual)
Dates: Start 2015-11-23 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Change in percentage of patients meeting the exercise goal | baseline, 3, 6, and 12 months]
  moderate exercise for ≥150 min/week or strenuous exercise for ≥75 min/week (* ≥12.5 MET-hr/week for lung cancer patients; no limit on exercise strength)
Change in percentage of patients meeting the body mass index (BMI) goal | baseline, 3, 6, and 12 months
  BMI in kg/m^2 goal 18.5-22.9 (≥18.5 for lung cancer patients)
Change in percentage of patients meeting the posttraumatic growth inventory (PTGI) goal | 3, 6, and 12 months
  General is a quality of life measure with higher scores indicating better quality of life (range 0-105)

SECONDARY OUTCOMES:
Change in percentage of patients meeting diet goal | baseline, 3, 6, and 12 months
  Mini Dietary assessment Index (MDI) score ≥ 80
Change in execution level of health habits | baseline, 3, 6, and 12 months
  10 Rules for Highly Effective Health Behavior
Change in level of anxiety and depression | baseline, 3, 6, and 12 months
  We measured psychologic distress with the Hospital Anxiety and Depression Scale (HADS), which consists of 14 items (7 for anxiety and 7 for depression).
Change in level of fatigue | baseline, 3, 6, and 12 months
  The Brief Fatigue Inventory (BFI) scale, which consists of 9 items that rate fatigue severity and interference on a 0-to-10 scale,
Change in level of self-management strategy | baseline, 3, 6, and 12 months
  We assessed the SM strategies of health with the SMASH Assessment Tool (SAT), which is a three-set, 16-factor, 91-item tool (i.e., the core strategies with 28 items, preparation strategies with 30 items, and implementation strategies with 33 items) that assesses the patients' ability to overcome their health-related crisis.
Change in level of social support and spiritual well-being | baseline, 3, 6, and 12 months
  The social support (2 items) and spiritual (6 items) scales of the McGill Quality of Life (McGill QOL)
Cost effectiveness analysis | baseline, 3, 6, and 12 months
  Cost effectiveness analysis

CONTACTS AND LOCATIONS:
Overall Officials: Young Ho Yun, MD. PhD, Principal Investigator — Seoul National University Hospital
Locations (4):
- South Korea (4):
  - Eun Sook Lee, Ilsan, Gyeonggi-do
  - Sung Kim, Seoul
  - Eun Mi Nam, Seoul
  - Kyung Hae Jung, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Ahlberg K, Ekman T, Gaston-Johansson F, Mock V. Assessment and management of cancer-related fatigue in adults. Lancet. 2003 Aug 23;362(9384):640-50. doi: 10.1016/S0140-6736(03)14186-4. PMID 12944066
- [Background] Andersson G, Bergstrom J, Hollandare F, Carlbring P, Kaldo V, Ekselius L. Internet-based self-help for depression: randomised controlled trial. Br J Psychiatry. 2005 Nov;187:456-61. doi: 10.1192/bjp.187.5.456. PMID 16260822
- [Background] Appel LJ, Clark JM, Yeh HC, Wang NY, Coughlin JW, Daumit G, Miller ER 3rd, Dalcin A, Jerome GJ, Geller S, Noronha G, Pozefsky T, Charleston J, Reynolds JB, Durkin N, Rubin RR, Louis TA, Brancati FL. Comparative effectiveness of weight-loss interventions in clinical practice. N Engl J Med. 2011 Nov 24;365(21):1959-68. doi: 10.1056/NEJMoa1108660. Epub 2011 Nov 15. PMID 22085317
- [Background] Barsevick AM, Dudley W, Beck S, Sweeney C, Whitmer K, Nail L. A randomized clinical trial of energy conservation for patients with cancer-related fatigue. Cancer. 2004 Mar 15;100(6):1302-10. doi: 10.1002/cncr.20111. PMID 15022300
- [Background] Brendryen H, Kraft P. Happy ending: a randomized controlled trial of a digital multi-media smoking cessation intervention. Addiction. 2008 Mar;103(3):478-84; discussion 485-6. doi: 10.1111/j.1360-0443.2007.02119.x. PMID 18269367
- [Background] Burton AW, Fanciullo GJ, Beasley RD, Fisch MJ. Chronic pain in the cancer survivor: a new frontier. Pain Med. 2007 Mar;8(2):189-98. doi: 10.1111/j.1526-4637.2006.00220.x. PMID 17305690
- [Background] Courneya KS, Friedenreich CM, Sela RA, Quinney HA, Rhodes RE, Handman M. The group psychotherapy and home-based physical exercise (group-hope) trial in cancer survivors: physical fitness and quality of life outcomes. Psychooncology. 2003 Jun;12(4):357-74. doi: 10.1002/pon.658. PMID 12748973
- [Background] Courneya KS, Mackey JR, Bell GJ, Jones LW, Field CJ, Fairey AS. Randomized controlled trial of exercise training in postmenopausal breast cancer survivors: cardiopulmonary and quality of life outcomes. J Clin Oncol. 2003 May 1;21(9):1660-8. doi: 10.1200/JCO.2003.04.093. PMID 12721239
- [Background] Daley AJ, Crank H, Saxton JM, Mutrie N, Coleman R, Roalfe A. Randomized trial of exercise therapy in women treated for breast cancer. J Clin Oncol. 2007 May 1;25(13):1713-21. doi: 10.1200/JCO.2006.09.5083. PMID 17470863
- [Background] Demark-Wahnefried W, Clipp EC, Lipkus IM, Lobach D, Snyder DC, Sloane R, Peterson B, Macri JM, Rock CL, McBride CM, Kraus WE. Main outcomes of the FRESH START trial: a sequentially tailored, diet and exercise mailed print intervention among breast and prostate cancer survivors. J Clin Oncol. 2007 Jul 1;25(19):2709-18. doi: 10.1200/JCO.2007.10.7094. PMID 17602076
- [Background] Morey MC, Snyder DC, Sloane R, Cohen HJ, Peterson B, Hartman TJ, Miller P, Mitchell DC, Demark-Wahnefried W. Effects of home-based diet and exercise on functional outcomes among older, overweight long-term cancer survivors: RENEW: a randomized controlled trial. JAMA. 2009 May 13;301(18):1883-91. doi: 10.1001/jama.2009.643. PMID 19436015
- [Background] Fawzy NW. A psychoeducational nursing intervention to enhance coping and affective state in newly diagnosed malignant melanoma patients. Cancer Nurs. 1995 Dec;18(6):427-38. PMID 8564938
- [Background] Gessler S, Low J, Daniells E, Williams R, Brough V, Tookman A, Jones L. Screening for distress in cancer patients: is the distress thermometer a valid measure in the UK and does it measure change over time? A prospective validation study. Psychooncology. 2008 Jun;17(6):538-47. doi: 10.1002/pon.1273. PMID 17973237
- [Background] Lachin JM. Sample size determinants for r X c comparative trials. Biometrics. 1977 Jun;33(2):315-24. No abstract available. PMID 884194
- [Background] Moher D, Schulz KF, Altman DG. The CONSORT statement: revised recommendations for improving the quality of reports of parallel-group randomised trials. Lancet. 2001 Apr 14;357(9263):1191-4. PMID 11323066
- [Background] Svetkey LP, Stevens VJ, Brantley PJ, Appel LJ, Hollis JF, Loria CM, Vollmer WM, Gullion CM, Funk K, Smith P, Samuel-Hodge C, Myers V, Lien LF, Laferriere D, Kennedy B, Jerome GJ, Heinith F, Harsha DW, Evans P, Erlinger TP, Dalcin AT, Coughlin J, Charleston J, Champagne CM, Bauck A, Ard JD, Aicher K; Weight Loss Maintenance Collaborative Research Group. Comparison of strategies for sustaining weight loss: the weight loss maintenance randomized controlled trial. JAMA. 2008 Mar 12;299(10):1139-48. doi: 10.1001/jama.299.10.1139. PMID 18334689
- [Background] Vallance JK, Courneya KS, Plotnikoff RC, Yasui Y, Mackey JR. Randomized controlled trial of the effects of print materials and step pedometers on physical activity and quality of life in breast cancer survivors. J Clin Oncol. 2007 Jun 10;25(17):2352-9. doi: 10.1200/JCO.2006.07.9988. PMID 17557948
- [Background] Yun YH, Lee MK, Bae Y, Shon EJ, Shin BR, Ko H, Lee ES, Noh DY, Lim JY, Kim S, Kim SY, Cho CH, Jung KH, Chun M, Lee SN, Park KH, Chang YJ. Efficacy of a training program for long-term disease- free cancer survivors as health partners: a randomized controlled trial in Korea. Asian Pac J Cancer Prev. 2013;14(12):7229-35. doi: 10.7314/apjcp.2013.14.12.7229. PMID 24460280
- [Background] Yun YH, Sim JA, Jung JY, Noh DY, Lee ES, Kim YW, Oh JH, Ro JS, Park SY, Park SJ, Cho KH, Chang YJ, Bae YM, Kim SY, Jung KH, Zo ZI, Lim JY, Lee SN. The association of self-leadership, health behaviors, and posttraumatic growth with health-related quality of life in patients with cancer. Psychooncology. 2014 Dec;23(12):1423-30. doi: 10.1002/pon.3582. Epub 2014 May 21. PMID 24844184
- [Background] Yun YH, Jung JY, Sim JA, Choi H, Lee JM, Noh DY, Han W, Park KJ, Jeong SY, Park JW, Wu HG, Chie EK, Kim HJ, Lee JH, Zo ZI, Kim S, Lee JE, Nam SJ, Lee ES, Oh JH, Kim YW, Kim YT, Shim YM. Patient-reported assessment of self-management strategies of health in cancer patients: development and validation of the Smart Management Strategy for Health Assessment Tool (SAT). Psychooncology. 2015 Dec;24(12):1723-30. doi: 10.1002/pon.3839. Epub 2015 May 26. PMID 26014043
- [Background] Hawkes AL, Chambers SK, Pakenham KI, Patrao TA, Baade PD, Lynch BM, Aitken JF, Meng X, Courneya KS. Effects of a telephone-delivered multiple health behavior change intervention (CanChange) on health and behavioral outcomes in survivors of colorectal cancer: a randomized controlled trial. J Clin Oncol. 2013 Jun 20;31(18):2313-21. doi: 10.1200/JCO.2012.45.5873. Epub 2013 May 20. PMID 23690410
- [Background] Katon WJ, Lin EH, Von Korff M, Ciechanowski P, Ludman EJ, Young B, Peterson D, Rutter CM, McGregor M, McCulloch D. Collaborative care for patients with depression and chronic illnesses. N Engl J Med. 2010 Dec 30;363(27):2611-20. doi: 10.1056/NEJMoa1003955. PMID 21190455